CLINICAL TRIAL: NCT03867760
Title: Efficacy and Mechanistic Testing of a Self-Management Intervention for Managing Chronic Pain With Cancer Survivors
Brief Title: Self-Management Interventions for Chronic Pain Relief With Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Linda Eaton, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004809; 5K23NR017208 (NIH); RG1004569 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-00201 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will use the recorded hypnosis intervention (RHI) at home for 28 days.
  Interventions: Behavioral: Recorded Hypnosis Intervention
- Attention Control Group (Active Comparator): Participants will use a recorded relaxation intervention at home for 28 days.
  Interventions: Behavioral: Recorded Relaxation Intervention

INTERVENTIONS:
Behavioral: Recorded Hypnosis Intervention — The RHI consists of four digital recordings developed by the investigator using standardized hypnosis scripts for pain reduction and uploaded to a MP3 player. The scripts were developed for patients with chronic pain and tested by a psychologist who is an expert in hypnosis research. Participants will listen to the recordings daily for 28 days in the prescribed order (4 recordings for 3 days each, and then any recording for the remaining 16 days). The script includes an induction, suggestions for how to access inner resources and manage pain, and post-hypnotic suggestions for permanence of hypnosis benefits and self-hypnosis practice.
  Arms: Intervention Group
Behavioral: Recorded Relaxation Intervention — The recorded relaxation intervention consists of four digital recordings developed by the investigator using standardized relaxation scripts and uploaded to a MP3 player. Participants will listen to the recordings daily for 28 days in the prescribed order (4 recordings for 3 days each, and then any recording for the remaining 16 days).
  Arms: Attention Control Group

SUMMARY:
Cancer survivors who suffer from chronic pain would benefit from a low-cost, self-management intervention they can use at home. This study will evaluate the efficacy of a recorded hypnosis intervention in reducing chronic pain among cancer survivors and will explore its biological and psychological mechanisms.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to evaluate if a 4-week recorded hypnosis intervention (RHI) works for reducing chronic pain in 100 adult cancer survivors who have completed active treatment. The RHI will be compared to an attention control condition (relaxation recording). qEEG measurement will be obtained while listening to the RHI at weeks 0, 2, and 4 to explore if brain states are related to hypnotic analgesia during the 4-week study period in 20 study participants.

The study has the following specific aims:

Aim 1: Does the RHI work? Evaluate the efficacy of RHI in reducing self-reported pain intensity (primary outcome), pain interference, anxiety, depression, fatigue and sleep disturbance (secondary outcomes) at 4 weeks compared to the attention control condition (relaxation recording). Hypothesis: RHI will significantly reduce pain intensity, pain interference, anxiety, depression, fatigue, and sleep disturbance at 4 weeks.

Aim 2: For whom does the RHI work? Examine if psychological factors (hypnotic suggestibility, mental absorption, treatment outcome expectancy, fear of cancer recurrence, resilience, self-efficacy) influence the relationship between RHI and pain intensity at weeks 0, 2, and 4.

Aim 3: How does the RHI work? a. Compare brain activity as measured by electroencephalogram (EEG) in cancer survivors with chronic pain (n=30) receiving the RHI relative to the attention control condition (relaxation recording) at weeks 0, 2, and 4. b. Explore the effects of brain activity on pain intensity at weeks 0, 2, and 4. In addition, structured interviews will be conducted with participants to understand facilitators and barriers associated with undergoing EEG at three time points and perceptions on how the intervention works to reduce pain.

ELIGIBILITY:
Inclusion Criteria:

* self-reporting moderate or higher pain on average during the last week (> 3 on a 0-10 pain intensity numeric scale)
* self-reporting experiencing pain at least half of the days in the past 4 weeks
* self-reporting chronic pain related to cancer or its treatment
* completed active cancer treatment other than maintenance therapy
* being > 18 years of age
* functional fluency in English
* mentally and physically able to participate and complete surveys

Exclusion Criteria:

• has a psychiatric condition or symptoms (i.e., diagnosis of paranoid schizophrenia or active paranoid delusional thoughts, as determined via a telephone or in-person screening assessment) that would interfere with study participation.

Exclusion Criteria for Optional EEG Measurement:

* a history of seizure condition within the last year
* a significant brain injury or skull defect
* a history of brain cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Eaton, RN, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from adult cancer survivors with chronic pain. The final data set will include (1) qEEG pattern data, and (2) self-reported demographic and behavioral data from questionnaires and interviews. The final data set will be stripped of individual identifiers prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8/31/21 - 8/31/24
Access Criteria: The data and associated documentation will be made available to users only under a data-sharing agreement that provides for (a) a commitment to using the data only for research purposes and not to identify any individual participant, (b) a commitment to securing the data using appropriate computer technology, and (c) a commitment to destroying or returning the data after analyses are completed. Such a data-use agreement will be executed through the PI. The database can then be accessed via a secure website, in a format that can be used by a variety of statistical software packages.

REFERENCES:
- [Derived] Eaton LH, Jang MK, Jensen MP, Pike KC, Heitkemper MM, Doorenbos AZ. Hypnosis and relaxation interventions for chronic pain management in cancer survivors: a randomized controlled trial. Support Care Cancer. 2022 Dec 17;31(1):50. doi: 10.1007/s00520-022-07498-1. PMID 36526937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by phone and during cancer survivor or palliative care clinic visits from February 2019 to August 2021.
Period: Overall Study
Arm/Group | Intervention Group | Attention Control Group
Started | 55 | 54
Completed | 49 | 46
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — subject could not meet study logistics | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Hypnosis: Participants were asked to use the recorded hypnosis intervention for 28 days.
- Relaxation: Participants were asked to use the recorded relaxation intervention for 28 days.
- Total: Total of all reporting groups
Arm/Group | Hypnosis | Relaxation | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.6) | 56.8 (12.2) | 55.62 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 89
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 16 | 24
  White | 35 | 35 | 70
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 4 | 2 | 6
Stanford Hypnotic Clinical Scale for Adults [Mean (Standard Deviation); unit: units on a scale] — The Stanford Hypnotic Clinical Scale for Adults involves a standard hypnotic induction followed by five standard hypnotic suggestions delivered by a member of the research team. Participant responses to the suggestions are coded (yes/no) and responses are summed to create the total scale score, which can range from 0 to 5. A higher score indicates a higher level of hypnotic responsivity.
  units on a scale | 2.78 (1.44) | 2.81 (1.39) | 2.80 (1.40)
Tellegen Absorption Scale [Mean (Standard Deviation); unit: units on a scale] — The 34-item multi-dimensional scale measures imaginative involvement and the tendency to become mentally absorbed in everyday activities. The minimum score is 0 and the maximum score is 34. A higher score indicates a higher level of mental absorption.
  units on a scale | 15.67 (7.78) | 14.52 (8.60) | 15.10 (8.18)
Credibility Expectancy Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Credibility Expectancy Questionnaire consists of 6 items using the 0 -10 numeric rating scale to measure ratings of beliefs about how well the treatment might reduce pain. Scores range from 0 to 60 with higher scores indicating greater belief in the treatment's effect in reducing their pain.
  units on a scale | 45.96 (24.55) | 55.33 (22.01) | 50.54 (23.69)
PROMIS®, v.1.0, 1a - Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Outcomes Measurement Information System® (PROMIS®) v.1.0, 1a - Pain Intensity: Average pain intensity was assessed by asking participants to rate their pain intensity on average in the past 7 days using the 0-10 numeric rating scale with 0 = "no pain" and 10 = "worst pain imaginable."
  units on a scale | 6.05 (1.83) | 6.02 (1.86) | 6.04 (1.84)
PROMIS®, Pain Interference SF4v1.1 [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System® (PROMIS®) Pain Interference Short Form 4v1.1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less pain interference.
  units on a scale | 61.62 (6.49) | 62.16 (6.58) | 61.89 (6.51)
PROMIS®, Anxiety SF4v1 [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System® (PROMIS®) Anxiety Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less anxiety.
  units on a scale | 59.53 (8.26) | 58.71 (9.53) | 59.13 (8.88)
PROMIS®, Depression SF4v1 [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System® (PROMIS®) Depression Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less depression.
  units on a scale | 53.89 (8.54) | 53.76 (8.90) | 53.82 (8.68)
PROMIS®, Fatigue SF4v1 [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System® (PROMIS®) Fatigue Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less fatigue.
  units on a scale | 58.01 (8.58) | 58.36 (9.44) | 58.18 (8.98)
PROMIS®, Sleep Disturbance SF4v1 [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System® (PROMIS®) Sleep Disturbance Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less sleep disturbance.
  units on a scale | 55.61 (7.52) | 54.36 (9.51) | 54.99 (8.55)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) v.1.0, 1a - Pain Intensity; minimum value 0, maximum value 10; a lower score indicates a better outcome. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: Cancer survivors with chronic pain were randomly assigned to the recorded hypnosis intervention group or the attention control group (recorded relaxation intervention).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Participants who use the recorded hypnosis intervention for 28 days.
- Attention Control Group: Participants who use the recorded relaxation intervention for 28 days.
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -1.61 (1.88) | -1.35 (1.54)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in pain intensity than cancer survivors assigned to the relaxation intervention; Test type: Superiority — The study was designed to detect a difference in pain intensity of at least 0.85 points corresponding to an effect size of 0.57 based on results from our pilot study. The sample size needed was 50 per group based on power of .80, alpha of .05; p = 0.809, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in addition to baseline pain medications in the ANCOVA analysis

2. Secondary Outcome: Change in Pain Interference
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) Pain Interference Short Form 4v1.1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less pain interference. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -3.75 (5.38) | -3.03 (6.81)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in pain interference than cancer survivors assigned to the relaxation intervention; Test type: Superiority; p = 0.369, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in addition to baseline pain medications in the ANCOVA analysis

3. Secondary Outcome: Change in Anxiety
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) Anxiety Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less anxiety. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -3.07 (6.11) | -3.61 (6.80)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in anxiety than cancer survivors assigned to the relaxation intervention; Test type: Superiority; p = 0.029, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in the ANCOVA analysis

4. Secondary Outcome: Change in Depression
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) Depression Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less depression. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -1.75 (5.35) | -2.74 (6.81)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in depression than cancer survivors assigned to the relaxation intervention; Test type: Superiority; p = 0.236, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in the ANCOVA analysis

5. Secondary Outcome: Change in Fatigue
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) Fatigue Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less fatigue. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -2.66 (5.65) | -2.67 (7.39)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in fatigue than cancer survivors assigned to the relaxation intervention; Test type: Superiority; p = 0.904, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in the ANCOVA analysis

6. Secondary Outcome: Change in Sleep Disturbance
Description: The Patient Reported Outcomes Measurement Information System® (PROMIS®) Sleep Disturbance Short Form 4v1 scores were converted to T-scores. T-scores of 50 indicates the U.S. population mean with a standard deviation of 10. A lower score indicates less sleep disturbance. A change between pre-treatment (baseline) and post-treatment (4 weeks) scores is reported.
Time Frame: Pre- to Post-treatment (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 49 | 46
score on a scale | -3.96 (7.34) | -3.31 (9.49)
Statistical Analysis 1: Comparison: Intervention Group vs Attention Control Group; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention for 28 days will not report significantly greater pre- to post-treatment decreases in sleep disturbance than cancer survivors assigned to the relaxation intervention; Test type: Superiority; p = 0.936, ANCOVA — An a priori significance level was set at 0.05; We controlled for pre-treatment scores in the ANCOVA analysis

7. Other Pre Specified Outcome: Treatment Credibility and Expectancy
Description: Credibility and Expectancy Questionnaire; minimum score = 0, maximum score = 60; a higher score indicates a better outcome. Pre-treatment (baseline) scores were calculated for hypnosis participants with a clinically meaningful improvement in pain intensity (change from pre-treatment to post-treatment of at least 2 points) and for hypnosis participants who did not have a clinically meaningful improvement in pain intensity.
Time Frame: Pre-treatment
Population: Cancer survivors with chronic pain who use the recorded hypnosis intervention for 28 days. Participants in the Attention Control Group were not assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Hypnosis Improvers: Hypnosis participants who experienced a clinically meaningful improvement in pain intensity (defined as experiencing at least a 2-point [0 - 10 numeric pain scale] reduction in pain intensity from pre- to post-treatment).
- Hypnosis Non-Improvers: Hypnosis participants who did not experience a clinically meaningful improvement in pain intensity (defined as experiencing at least a 2-point [0 - 10 numeric pain scale] reduction in pain intensity from pre- to post-treatment).
Arm/Group | Hypnosis Improvers | Hypnosis Non-Improvers
Number analyzed (Participants) | 27 | 22
score on a scale | 53.81 (23.55) | 36 (24.7)
Statistical Analysis 1: Comparison: Hypnosis Improvers; Null Hypothesis: Cancer survivors with chronic pain assigned to the daily use of the hypnosis intervention who experience a clinically meaningful improvement in pain intensity will not have a significantly higher pre-treatment treatment credibility and expectancy score than non-improvers; Test type: Superiority; p = 0.02, t-test, 2 sided — An a priori significance level was set at 0.05

8. Other Pre Specified Outcome: Change in Brain Activity
Description: EEG measurement; measures brain activity while using study intervention. Participants underwent an EEG while listening to the assigned study intervention at three time points: pre-treatment (baseline), mid-treatment (2 weeks), and post-treatment (4 weeks).
Time Frame: Baseline, 2 weeks, 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to post-treatment (4 weeks)
Groups:
- Intervention Group: Participants are asked to use the recorded hypnosis intervention for 28 days.
- Attention Control Group: Participants are asked to use a recorded relaxation intervention for 28 days.
Arm/Group | Intervention Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

LIMITATIONS AND CAVEATS:
We were unable to conduct EEGs throughout the study period due to restrictions at the data collection site during the COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03867760/Prot_SAP_001.pdf